CLINICAL TRIAL: NCT01473251
Title: Analysis of Growth Factors in Patients Undergoing Lucentis or Avastin Injections for Diabetic Macular Edema and Exudative Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitreo-Retinal Associates, Michigan (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VARI 2011 002
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Exudative Macular Degeneration; Diabetic Macular Edema
MeSH Terms: conditions — Wet Macular Degeneration | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Avastin for Diabetic Macular Edema (Active Comparator): 1.25 mg avastin monthly for 4 months
  Interventions: Drug: Avastin
- Avastin for Exudative Macular Degeneration (Active Comparator): 1.25 mg Avastin monthly for 4 months
  Interventions: Drug: Avastin
- Lucentis for Exudative Macular Degeneration (Active Comparator): 0.5 mg Lucentis monthly for 4 months
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Avastin — 1.25 mg monthly for 4 months
  Arms: Avastin for Diabetic Macular Edema
Drug: Avastin — 1.25 mg monthly for 4 months
  Arms: Avastin for Exudative Macular Degeneration
Drug: Lucentis — 0.5 mg monthly for 4 months
  Arms: Lucentis for Exudative Macular Degeneration

SUMMARY:
The purpose of this study is to measure biomarkers in the vitreous of patients undergoing Lucentis or avastin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 85 with diabetes and hemoglobin A1C </= 10, or exudative macular degeneration.
* Diabetic macular edema with average retinal thickness central subfield >/= 290um.

Exclusion Criteria:

* Macular atrophy/fibrosis.
* Ocular anti-VEGF treatment within 3 months.
* Treatment with topical or oral carbonic-anhydrase inhibitor within one month
* Laser photocoagulation within 3 months (diabetic cohort)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Analysis of collected vitreous samples to identify biomarkers. | End of study
  Analysis of collected vitreous samples in regards to identification of biomarkers that are prognostic for response to anti-angiogenic treatment of retinopathy, and the exploration of a more effective dosing regiment for intravitreal injections of Lucentis/Avastin for exudative macular degeneration and Avastin for diabetic macular edema.

CONTACTS AND LOCATIONS:
Overall Officials: Louis C. Glazer, MD, Principal Investigator — Vitreo Retinal Associates
Locations (1):
- Vitreo-Retinal Associates, Grand Rapids, Michigan, United States